CLINICAL TRIAL: NCT02551263
Title: Prospective Observational Study to Explore the Efficacy of Eribulin as 1st-line or 2nd-line Chemotherapy in Patients With HER2-negative Hormone-resistant Inoperable or Recurrent Metastatic Breast Cancer
Brief Title: Eribulin Treatment as 1st-line or 2nd-line Chemotherapy for HER2-negative Hormone-resistant Inoperable or Recurrent Metastatic Breast Cancer
Acronym: E-SPEC
Status: Completed | Type: Observational
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Kyoto Breast Cancer Research Network (Other)
Responsible Party: Sponsor
Other Study IDs: TRIBC1505; UMIN000018178 (Registry Identifier: UMIN-CTR)
Record Dates: First submitted 2015-09-15; First posted 2015-09-16 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Eribulin; HER2-negative; hormone-resistant; inoperable; recurrent metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — eribulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational group: All patients will receive adequate treatment for breast cancer which selected by the primary physician after enrollment using the Japanese Breast Cancer Society Clinical Practice Guideline of Breast Cancer and the National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines in Oncology. Investigators at the investigational sites will enter patient data into an electronic data capture (EDC) system up to the third chemotherapy in the study.
  Interventions: Drug: Eribulin

INTERVENTIONS:
Drug: Eribulin — Eribulin 1.4 mg/m2 will be administered intravenously over 2 to 5 minutes on day 1 and 8 of every 21-day cycle, in a real-world setting.

SUMMARY:
This is a observational study in a real-world setting, not requiring determining a dosage regimen, dose reduction criteria, rest period criteria and withdrawal criteria. The purpose of the study is to investigate the efficacy of eribulin as the first or second line chemotherapy to prolong overall survival and to explore factors affecting the survival in patients with HER2-negative hormone-resistant inoperable or recurrent metastatic breast cancer who scheduled to receive the first or second line chemotherapy in clinical practice in Japan. The total duration of the study will be a maximum of 5 years, consisting of 2-year enrollment period and 3-year observational period; the duration of patient participation will be 3 years. All patients will receive adequate treatment for breast cancer which selected by the primary physician after enrollment using the Japanese Breast Cancer Society Clinical Practice Guideline of Breast Cancer and the National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines in Oncology. Investigators at the investigational sites will enter patient data into an electronic data capture (EDC) system up to the third chemotherapy in the study. The end of the study is defined as the time the last patient completes observational period. Patients will primarily be assessed by overall survival (OS) of the first line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with histologically or cytologically confirmed breast cancer.
2. Patients with inoperable or recurrent metastatic breast cancer regardless of the metastatic site and number, excluding symptomatic central nervous system metastases.
3. Patients with HER2-negative disease confirmed as ISH negative or IHC 0, 1+ or 2+ (Those with IHC 2+ are eligible, if the additional ISH test results are negative. Those are ineligible who are with any positive results of estrogen receptor or progesterone receptor test on primary and recurrent lesion).
4. Patients who are resistant to hormone therapy.
5. Patients with indication for the first or second line chemotherapy in HER2-negative hormone-resistant inoperable or recurrent metastatic breast cancer who are scheduled to receive the chemotherapy.
6. Patients with the Eastern Cooperative Oncology Group (ECOG) performance status score 0-3 at the time of enrollment.
7. Patients with adequate bone marrow and major organ function judged by the primary physician.
8. Patients who have signed written informed consent to participate in this study.

Exclusion Criteria:

1. Patients with symptomatic metastasis in the central nervous system.
2. Patients with a previous history of hypersensitivity to any component of drugs which will be administered in the treatment.
3. Patients who are considered to be inappropriate for the study participation by the primary physician.

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with HER2-negative hormone-resistant inoperable or recurrent metastatic breast cancer, who are scheduled to receive the first or second line chemotherapy in clinical practice in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2015-07-22 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) of the first line chemotherapy | From starting date of the first line chemotherapy until date of death from any cause (up to 5 years)

SECONDARY OUTCOMES:
Overall survival (OS) of the second and third line chemotherapy | From starting date of each line of chemotherapy until date of death from any cause (up to 5 years)
Progression-free survival (PFS) of the first, second and third line chemotherapy | From starting date of each line of chemotherapy until the date of first documented disease progression or date of death from any cause, whichever comes first (up to 5 years)
Post progression survival (PPS) of the first, second and third line chemotherapy | From the date of first documented disease progression in each line of chemotherapy until date of death from any cause (up to 5 years)
Time to treatment failure (TTF) of the first, second and third line chemotherapy | From starting date of each line of chemotherapy until date of discontinuation of study treatment for any reason including disease progression, treatment toxicity or death (up to 5 years)
New metastasis-free survival (nMFS) of the first, second and third line chemotherapy | From starting date of each line of chemotherapy until the date of first documented disease progression due to appearance of a new metastasis or date of death from any cause, whichever comes first (up to 5 years)
Assessment and comparison of Quality Adjusted Life Years (QALYs) in the first, second and third line chemotherapy, using Japanese version of the EQ-5D-5L value set | From date of the baseline QALYs assessment in each line of chemotherapy until the last date of each line of chemotherapy (up to 5 years)
Serious adverse events | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yuichiro Kikawa, MD, Principal Investigator — Kobe City Medical Center General Hospital; Takeshi Kotake, MD, Principal Investigator — Kyoto University
Locations (2):
- Japan (2):
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kyoto University Hospital, Kyoto, Kyoto